CLINICAL TRIAL: NCT02232451
Title: Comparison of Loop-tip Cook Medical® Wire vs Traditional Endoscopic Technique Cannulation in the Prevention of Post-ercp Pancreatitis and Biliary Tree Access in High-risk Patients
Brief Title: Comparison of Loop-tip Cook Medical® Wire Versus Traditional Endoscopic Technique
Acronym: loop
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliera San Paolo (Other)
Responsible Party: Principal Investigator, Enzo Masci, Chief of Gastrointestinal Endoscopy, Azienda Ospedaliera San Paolo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: loop20216
Record Dates: First submitted 2012-08-01; First posted 2014-09-05 (Estimated); Last update posted 2014-09-25 (Estimated); Status verified 2014-09

CONDITIONS: Complications of Surgical and Medical Care: General Terms
Keywords: loop; ERCP; cannulation; biliary; wire
MeSH Terms: interventions — Cholangiopancreatography, Endoscopic Retrograde; Catheterization

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ERCP with loop tip wire (Experimental): ERCP with loop tip wire is an endoscopic procedure to treat biliary disease. Wire guide cannulation with loop-tip is a new procedure to improve rate of biliary cannulation and reduce complication, as post-procedure pancreatitis.
  Interventions: Device: ERCP with loop tip wire
- ERCP for cannulation (Active Comparator): ERCP for cannulation of CBD with traditional technique
  Interventions: Device: ERCP for cannulation

INTERVENTIONS:
Device: ERCP with loop tip wire — Endoscopic retrograde cholangio-pancreatography with guide wire (loop-tip) for CBD cannulation
  Arms: ERCP with loop tip wire
Device: ERCP for cannulation — Endoscopic retrograde cholangio-pancreatography with traditional technique for CBD cannulation
  Arms: ERCP for cannulation

SUMMARY:
The purpose of this study is to test a new guide-wire (loop-tip wire) with a loop in the tip for the prevention of PEP and biliary tree access, in post-ERCP pancreatitis in high-risk patients.

DETAILED DESCRIPTION:
Selective cannulation of common bile duct (CBD) by insertion of a guide-wire seems to be associated with fewer complication and post-ERCP pancreatitis (PEP) rate than the conventional biliary tree access with contrast injection even if results are conflicting. The aim of our study is to test a new guide-wire (loop-tip wire) with a loop in the tip for the prevention of PEP and biliary tree access, in PEP high-risk patients.

Type of study: Multicentric, prospective and randomized trial

Patients: PEP high-risk patients underwent ERCP for benign biliary pathology

Number of patients: 320 patients (160 for each group)

Aim:

Primary end point: The evaluation of the incidence of PEP . Secondary end point: The evaluation of CBD percentage cannulation.

ELIGIBILITY:
Inclusion Criteria:

* high risk patients for post-ERCP pancreatitis

Exclusion Criteria:

* age < 18 yrs
* allergy to the contrast medium
* previous surgery
* neoplastic bilio-pancreatic disease
* previous EBS

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Actual)
Dates: Start 2010-11; Primary Completion 2012-06 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
The evaluation of the incidence of PEP | loop20216

SECONDARY OUTCOMES:
The evaluation of CBD percentage cannulation. | loop20216

CONTACTS AND LOCATIONS:
Overall Officials: Enzo Masci, MD, Study Director — Hospital San Paolo